CLINICAL TRIAL: NCT00463775
Title: Topiramate for Treatment of Patients With Borderline Personality Disorder and Alcohol Dependence
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment not progressing as planned.
Sponsor: Elizabeth Ralevski (Other)
Responsible Party: Sponsor-Investigator, Elizabeth Ralevski, Assistant Professor, Yale University
Organization: Yale University (Other)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 0702002346; ER0001
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Alcohol Dependence; Borderline Personality Disorder
Keywords: Treatment; Topiramate; Alcohol Dependence; Borderline Personality Disorder
MeSH Terms: conditions — Alcoholism; Borderline Personality Disorder | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Topiramate — SSRI plus topiramate SSRI plus placebo

SUMMARY:
The objective of the present study is to evaluate the efficacy of topiramate (250mg/day) versus placebo in decreasing aggression and reducing alcohol consumption in patients with borderline personality disorder (BPD) and alcohol dependence (AD).

DETAILED DESCRIPTION:
Background: Borderline personality disorder (BPD) affects about 2% of the American adult population. It is a very serious psychiatric disorder that places heavy demands on mental health resources. Behavior dysregulation (impulsivity, self-injurious acts, drinking or aggressive behavior) is considered one of the main features of BPD and is associated with significant clinical morbidity. Alcohol abuse is common among patients with BPD, and the co-morbid rates of alcoholism in BPD patients are estimated to be 30%. It has been hypothesized that alcohol misuse may be a manifestation of BPD's behavioral dysregulation. Also, BPD and alcohol dependence (AD) share a common underlying neurobiology. The co-occurrence of these disorders has been associated with increased rates of alcohol relapse, impulsive behaviors, greater resistance to treatment, and suicidal behavior. Effective treatment for patients with BPD and AD would result in markedly reduced health care costs and a substantial reduction in human distress and suffering. Despite dramatic advances in the treatment of BPD, to date, no single medication or types of medications have been uniquely identified as effective in treating BPD. Studies treating patients with co-morbid BPD and AD are expressly lacking.

Research Design and Methodology: This is an 8-week double-blind outpatient clinical trial of oral topiramate (250mg) vs placebo in individuals with BPD and AD. The study will be conducted at the West Haven, CT VA. Thirty men and women with a current diagnosis of BPD and AD will be enrolled. The State-Trait Anger Expression Inventory (STAEI) will be used to assess 5 aspects of aggression: state anger, trait anger, anger expressed inwardly, anger expressed outwardly, and anger control before and during treatment (weeks 0-8). The Timeline Follow-Back (TLFB) method will be used to document the degree of daily alcohol consumption before and during treatment (90 days before treatment, and weeks 0 - 8). Emergent side effects will be assessed using the modified version of the Systematic Assessment for Treatment Emergent Events (SAFTEE).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AD
* Diagnosis of BPD

Exclusion Criteria:

* Serious or unstable medical condition
* Opiate dependence
* Major Axis I disorder (bipolar disorder, schizophrenia)
* Taking mood stabilizers and antipsychotic medications
* LFT abnormalities that do not exceed 3 times normal values

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2007-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
drinking - measured using the TLFB | 12 weeks
craving - measured using the OCDS | 12 weeks
aggression - measured using the STAE | 12 weeks

SECONDARY OUTCOMES:
affect - measured using the Buss-Durkee Scale and Affective Intensity Scale | 12 weeks
side effects - measured using the SAFTEE | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Ralevski, Ph.D., Principal Investigator — Yale University

REFERENCES:
- [Derived] Stoffers-Winterling JM, Storebo OJ, Pereira Ribeiro J, Kongerslev MT, Vollm BA, Mattivi JT, Faltinsen E, Todorovac A, Jorgensen MS, Callesen HE, Sales CP, Schaug JP, Simonsen E, Lieb K. Pharmacological interventions for people with borderline personality disorder. Cochrane Database Syst Rev. 2022 Nov 14;11(11):CD012956. doi: 10.1002/14651858.CD012956.pub2. PMID 36375174